CLINICAL TRIAL: NCT02907814
Title: Objective, Prospective Measurement of Anterior Chamber Cell Grading Using Anterior Chamber Ocular Coherence Tomography
Brief Title: Measurement of Anterior Chamber Cell Grading Using Ocular Coherence Tomography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of administrative support
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, David S. Chu, MD, Clinical Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro20160000585
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Uveitis
Keywords: Uveitis; Optical Coherence Tomography
MeSH Terms: conditions — Uveitis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uveitis and Cataract Imaging Group (Experimental): Subjects will undergo up to three optical coherence tomography scans.
  Interventions: Device: Optical Coherence Tomography (OCT)
- Control (Experimental): Control subjects will undergo a brief, non-contact eye exam and then undergo up to three optical coherence tomography scans.
  Interventions: Device: Optical Coherence Tomography (OCT); Other: Eye Exam

INTERVENTIONS:
Device: Optical Coherence Tomography (OCT) — The OCT scan is a brief, non-contact scan of the back of the eye using infrared light. Subjects will see a light and be asked to look forwards while the scan is completed.
Other: Eye Exam — This is a brief, non-contact ocular exam.
  Arms: Control

SUMMARY:
Optical Coherence Tomography (OCT) is routinely used in ophthalmic clinical practice. It uses infrared light to image patient's eyes. Some patients, such as those with an inflammatory disease called uveitis or those who have just undergone cataract surgery, have intraocular inflammation. This intraocular inflammation commonly manifests as cells that can be seen on routine microscopic clinical examination. However, the only currently available method to quantify this intraocular inflammation is by manually counting on the microscopic clinical examination. The investigators plan to use the OCT machine to image patient's eyes. The investigators will then use the images obtained from the OCT to objectively quantify the degree of intraocular inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Intervention Arm:

  * Active anterior chamber inflammation in at least one eye as diagnosed by clinical exam
  * One of the following: 1) diagnosis of uveitis OR 2) undergone cataract extraction surgery within the previous 30 days
* Control Arm:

  * No active intraocular inflammation based on clinical exam

Exclusion Criteria:

* Corneal opacities in the affected eye
* Anyone judged unable to understand or consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Chu, MD, Principal Investigator — Rutgers University
Locations (1):
- Doctors Office Center, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempen JH, Ganesh SK, Sangwan VS, Rathinam SR. Interobserver agreement in grading activity and site of inflammation in eyes of patients with uveitis. Am J Ophthalmol. 2008 Dec;146(6):813-8.e1. doi: 10.1016/j.ajo.2008.06.004. Epub 2008 Aug 8. PMID 18687418
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] User Manual: SPECTRALIS HRA+OCT. Heidelberg Engineering GmbH;2012.
- [Background] Agarwal A, Ashokkumar D, Jacob S, Agarwal A, Saravanan Y. High-speed optical coherence tomography for imaging anterior chamber inflammatory reaction in uveitis: clinical correlation and grading. Am J Ophthalmol. 2009 Mar;147(3):413-416.e3. doi: 10.1016/j.ajo.2008.09.024. Epub 2008 Dec 3. PMID 19054493
- [Background] Li Y, Lowder C, Zhang X, Huang D. Anterior chamber cell grading by optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 Jan 9;54(1):258-65. doi: 10.1167/iovs.12-10477. PMID 23249705
- [Background] Igbre AO, Rico MC, Garg SJ. High-speed optical coherence tomography as a reliable adjuvant tool to grade ocular anterior chamber inflammation. Retina. 2014 Mar;34(3):504-8. doi: 10.1097/IAE.0b013e31829f73bd. PMID 23945636
- [Background] Sharma S, Lowder CY, Vasanji A, Baynes K, Kaiser PK, Srivastava SK. Automated Analysis of Anterior Chamber Inflammation by Spectral-Domain Optical Coherence Tomography. Ophthalmology. 2015 Jul;122(7):1464-70. doi: 10.1016/j.ophtha.2015.02.032. Epub 2015 Apr 4. PMID 25846846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ophthalmology clinic, Newark, New Jersey, from 10/26/2016 to 4/1/2018
Period: Overall Study
Arm/Group | Uveitis and Cataract Imaging Group | Control
Started | 6 | 0
Completed | 0 | 0
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Population: 6 subjects with uveitis identified in clinic and enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Uveitis and Cataract Imaging Group | Control | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12.5) |  | 40 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 2 |  | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 |  | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Identified Inflammatory Cells on OCT Scan
Description: This measure pertains to the identification of cells in OCT scan of the participants. The inflammatory cells to be identified refer to white blood cells. The anterior segment OCT scan was used to attempt to identify these cells in the anterior chamber of the eyes of the participants.
Time Frame: Through study completion, up to 1 year.
Population: Patients with uveitis identified from clinic.
Measure: Count of Participants; unit: Participants
Arm/Group | Uveitis and Cataract Imaging Group | Control
Number analyzed (Participants) | 6 | 0
Participants | 6 |

2. Secondary Outcome: Change in Cell Density Identified by OCT Scans Over Time
Description: Identification of changes in cell density in OCT scans over time
Time Frame: Baseline and up to 8 weeks.
Population: 0 of 6 patients had follow up data, unable to identify change over time.
Arm/Group | Uveitis and Cataract Imaging Group | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: entire study period, almost 2 years.
Arm/Group | Uveitis and Cataract Imaging Group | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0

LIMITATIONS AND CAVEATS:
Insufficient enrollment and follow up leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT02907814/Prot_SAP_000.pdf
  • Informed Consent Form (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02907814/ICF_001.pdf